CLINICAL TRIAL: NCT03994146
Title: Remifentanil Tapering and Post-adenotonsillectomy Pain in Children: a Randomised, Placebo Controlled, Double Blind Study
Brief Title: Remifentanil Tapering and Post-adenotonsillectomy Pain in Children
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Recruitment rate was not compatible with study completion
Sponsor: University Hospital, Akershus (Other)
Responsible Party: Principal Investigator, William James Morton, Principle Investigator, University Hospital, Akershus
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2019-001677-81
Record Dates: First submitted 2019-06-13; First posted 2019-06-21 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2023-08

CONDITIONS: Child, Only; Pain; Tonsillectomy; Remifentanil
MeSH Terms: conditions — Pain | interventions — Remifentanil; Sodium Chloride; Saline Solution

STUDY DESIGN:
Intervention Model Description: Double blind, randomised, placebo controlled trial.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Two syringes will be simultaneously infused during the operation. One will contain normal saline solution and the other remifentanil solution. Prior to the end of the operation one of the syringes will have a step wise decrease in infusion rate whilst the other will be abruptly stopped at the end of surgery.
  The syringes will be prepared according to randomisation in the hospital pharmacy and the identity of each syringe will be masked from all those involved in the study. The syringe randomisation will be de-coded following completion of recruitment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Remifentanil tapering / Placebo abrupt cessation (Experimental): Syringe one contains Remifentanil 2 mg in 40 ml NaCl 9 mg.ml-1 = 50 µg.ml-1 which will be infused at a rate of 0.9 µg.kg-1.min-1 and Syringe two contains 40 ml NaCl 9 mg.ml-1 at an identical infusion rate. According to randomisation syringe one will then be tapered towards the end of surgery and syringe two abruptly stopped.
  Interventions: Drug: Remifentanil; Drug: Sodium Chloride 9mg/mL
- Placebo tapering / Remifentanil abrupt cessation. (Placebo Comparator): Syringe one contains 40 ml NaCl 9 mg.ml-1 and Syringe two contains Remifentanil 2 mg in 40 ml NaCl 9 mg.ml-1 = 50 µg.ml-1 which will be infused at a rate of 0.9 µg.kg-1.min-1. According to randomization syringe one will be tapered towards the end of surgery and syringe two abruptly stopped.
  Interventions: Drug: Remifentanil; Drug: Sodium Chloride 9mg/mL

INTERVENTIONS:
Drug: Remifentanil — Syringe containing 40 ml of Remifentanil 50 µg/ml for intravenous administration.
  In order to maintain double blinding two identical syringes, prepared by pharmacy according to randomisation, will be simultaneously infused. One of the syringes will be abruptly stopped at the end of the operation whilst the other is tapered by stepwise decreases in infusion rate prior to the end of surgery.
  Other Names: Ultiva
Drug: Sodium Chloride 9mg/mL — Syringe containing 40 ml of Sodium Chloride 9 mg/ml for intravenous administration.
  In order to maintain double blinding two identical syringes, prepared by pharmacy according to randomisation, will be simultaneously infused. One of the syringes will be abruptly stopped at the end of the operation whilst the other is tapered by stepwise decreases in infusion rate prior to the end of surgery.
  Other Names: Normal saline; Placebo

SUMMARY:
Tonsillectomy is the commonest operation of childhood and results in considerable pain.

Remifentanil is a potent, ultra short acting opioid with a long- established safety record in paediatric anaesthesia that is used to provide intraoperative analgesia.

There is evidence from adult studies that remifentanil increases postoperative pain, although this may be ablated if propofol (rather than inhalational anaesthesia) is used or if the remifentanil is tapered rather than abruptly discontinued at the end of surgery.

The analgesic effect of gradual withdrawal of remifentanil at the end of surgery has not been studied in children and may have significant clinical implications.

The primary measure of efficacy will be the dose of fentanyl rescue analgesia in the peri-operative period (1 mcg.kg-1 bolus for >20% increase in pulse, blood pressure or movement intraoperatively or a FLACC(Face, Legs, Arms, Cry, Consolablity) score of >5 in recovery).

DETAILED DESCRIPTION:
Tonsillectomy is one of the commonest childhood operations in the world; approximately 9200 children have their tonsils removed every year in Norway alone.

Postoperative pain following the procedure is significant and notoriously difficult to mange. It´s management is potentially complicated by nausea and the risk of tonsillar infection or re-bleeding. Post-tonsillectomy pain in children is persistent, with 75% of children experiencing significant pain for the first three days and 50% still suffering with significant pain one week after the procedure. As well as delaying recovery, reducing oral intake of food and drink and disturbing sleep, post tonsillectomy pain has been shown to result in more than 50% of patients and their parents consulting their primary care physician in the post operative period, with the ensuing costs to the families and healthcare providers.

It is worth noting, that despite significant postoperative pain and potential complications, recovery after adeno / tonsillectomy is excellent.

The operative nature of tonsillectomy and adenotonsillectomy necessitates the provision of general anaesthesia to the child. The technique must ensure sufficient depth of anaesthesia and analgesia and protection of the airway from blood and surgical debris. Whilst there are a wide variety of anaesthetic techniques employed to achieve these goals,Total Intra Venous Anaesthesia (TIVA) with propofol and remifentanil has been shown in previous studies to be superior to volatile based (gas) anaesthesia, resulting in less post operative nausea and vomiting, less long term adverse behavioural changes, improved quality of emergence from anaesthesia, and less environmental pollution.

The use of remifentanil and propofol TIVA in children is well established and has been in use since at least the year 2000 for children undergoing tonsillectomy. Despite this the effects of remifentanil dosing on post-operative pain has not been studied in children undergoing tonsillectomy, though it may play a significant role.

ELIGIBILITY:
Inclusion Criteria:

* American Society Anaesthesiology I-II children 1 to 10 years
* Weight over 10.0 Kg
* Presenting for tonsillotomy / tonsillectomy or adenotonsillectomy at Akershus Universitetssykehus, Lørenskog and Lovisenberg Diakonale Hospital, Norway

Exclusion Criteria:

* Children who have had airway surgery previously.
* Children who have had any type of surgery in the previous 12 months.
* Children using chronic pain medication or who have used analgesia in the 24 hours preceding surgery.
* Children who are known to suffer from NSAID sensitive asthma.
* Children with a known allergy to propofol or remifentanil.
* Pre-existing cardiac, renal, liver dysfunction.
* Children or parents who are not fluent in Norwegian or English.
* Children in whom more than three attempts at intravenous cannulation are required or in those who request an inhalational induction or premedication

Ages: 1 Year to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 6 (Actual)
Dates: Start 2020-01-16 (Actual); Primary Completion 2023-08-18 (Actual); Study Completion 2023-08-18 (Actual)

PRIMARY OUTCOMES:
Intravenous fentanyl consumption in the perioperative period (mcg/kg). | From the induction of anaesthesia until discharge from the day case surgical unit.4 hours.
  Intravenous fentanyl consumption in the perioperative period (mcg/kg).

SECONDARY OUTCOMES:
Faces Legs Activity Cry Consolability (FLACC) pain scores at 20,40,60,90 and 120 minutes after the operation to give a Sum of Pain Intensity Differences (SPID). | From cessation of anaesthesia until 120 minutes after the cessation of anaesthesia.
  The Face, Legs, Activity, Cry, Consolability scale or FLACC scale is a well validated measurement used to assess pain for children or individuals that are unable to communicate their pain. The scale is scored in a range of 0-10 with 0 representing no pain. The scale has five criteria, which are each assigned a score of 0, 1 or 2.
  Thus the face component is scored as 0 for no particular expression or smile, 1 for an occasional grimace and 2 for a constant quivering chin or clenched jaw.
  The 0-2 score from each of the 5 domains is summated to give a total score between 0 and 10.
  A lower pain score indicates a better outcome than a high pain score.
Parents' Post Operative Pain Measure (PPOMP) on post operative days 1,3,7,10,14 and 28 | From the cessation of anaesthesia until the 28th day following discharge from the day case surgical unit.
  The Parents' Post Operative Pain Measure (PPOMP) is a well validated 15 point questionnaire used to measure childrens' pain after moderately or severely painful procedures.
  The parents are asked to complete the survey between particular times each day (e.g between supper and bed time). The questionnaire consists of 15 YES / NO questions such as: "When your child was recovering from surgery between supper and bed time today did s/he...
  Cry more easily than usual ? YES / NO
  Refuse to eat? YES/ NO
  Want to be closer to you than usual? YES / NO.
  The YES response are scored as 1 and the NO responses scores as 0. The sum score ranges from 0 to 15.
  A lower pain score indicates a better outcome than a high pain score.

CONTACTS AND LOCATIONS:
Overall Officials: Signe Søvik, MD. PhD, Principal Investigator — University Hospital, Akershus
Locations (2):
- Norway (2):
  - Akershsus Universitetssykehus, Lørenskog, Akershus
  - Lovisenberg Diakonale Sykehus, Oslo

IPD SHARING:
Plan to Share IPD: Yes
On request and following consultation with the Regional Ethics Committee and the Data Protection Officer at the host institution.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The data will be available following completion of the study and analysis and publication by the investigating team.
  There is no plan to time limit access to the data following this.
Access Criteria: On request and following consultation with the Regional Ethics Committee and the Data Protection Officer at the host institution.